CLINICAL TRIAL: NCT04101552
Title: Clinical and Radiographic Assessment of Immediate Implant Placement in Maxillary Esthetic Zone Using Socket Shield Technique With and Without the Use of Xenograft Particulate Graft Material
Brief Title: Investigate New Surgical Techniques to Improve Esthetics and Patient Satisfaction at Implant Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Poosy Hany Zaki Mohamed, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-6-3-2
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Fractured Tooth
MeSH Terms: conditions — Tooth Fractures | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- grafted versus graft less socket shield technique (Experimental)
  Interventions: Procedure: socket shield technique with xenophobic graft particulate and without the use of graft

INTERVENTIONS:
Procedure: socket shield technique with xenophobic graft particulate and without the use of graft — the jumping gap between the implant and the shield is grafted by xenograft particulate and the control group is not grafted

SUMMARY:
Many techniques have been proposed to prevent or rather minimize the labial bone resorption following extraction including guided bone regeneration techniques that has been attempted for many years now to preserve the alveolar ridge dimensions .

Immediate implant placement, flapless implant placement, palataly positioned implants and even platform switching.

However none of these methods were able to completely preserve the coronal part of the facial bone wall, and since the main reason of bone loss following extraction is the loss of the periodontal ligament, it seemed logical that root retention may affect the resorption process,The reason the root retention technique works in its different applications is due to the maintenance of the periodontal attachment including cementum, periodontal ligaments and bundle bone, this principle was used by Hurzeler in 2010 in a technique called socket shied technique.

DETAILED DESCRIPTION:
* The selected patients will be informed of the nature of the research work and informed consent will be obtained then randomized in equal proportions between control group conventional immediate implant placement with immediate temporization and study group socket shield technique with immediate temporization.
* Patients of both groups will be subjected to CBCT (diagnostic for upper arch).
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine)
* Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
* In the study group: along surgical fissure bur will be used for hemisectioning.
* The palatal portion will be carefully separated and extracted by a periotome and forceps.
* The osteomy site will be inspected and cleaned from any granulation tissue and the implant will be placed palatal to the tooth fragment.
* The jump gap was grafted with a xenogeneic bone particulate (De-proteinized bovine bone mineral Small granules (0.25-1 mm), the implant gained primary stability from bone apical and palatal sufficient to immediately restore with provisional restoration.
* In the control group: the root was hemisected using a fissure bur in a mesio-distal direction, and a traumatic removal of the palatal fragment of the root was achieved (no pressure was applied on it), then the buccal fragment was reduced using surgical bur leaving a thin layer of the root aspect intact to the buccal plate of the bone.
* The implant is placed in the socket in a way leaving space away from the remaining buccal plate without grafting this jumping gap
* The provisional restorations were relieved of occlusal contacts in centric occlusion and excursive movements. These restorations remained in situ for at least 6 to 12 weeks prior to any modifications or commencement of definitive restorative therapy
* A soft diet was recommended for the duration of the implant-healing phase. The patient was advised against functioning or activities to the implant site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable maxillary anterior teeth in the esthetic zone indicated for implant placement.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Uncontrolled diabetic patients.
* Pregnant patients.
* Teeth with Large pulpal pathosis as cysts, large periapical granulomas
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.
* Immunodeficiency pathology, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.
* Psychiatric problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | • Amount of bone loss will be measured after 6 month using linear measurement from CBCT
  Will be measured using linear measurements from CBCT

SECONDARY OUTCOMES:
secondary stability | will be measured intraoperative and 3 months after surgery
  Will be measured using Osstell

OTHER OUTCOMES:
pink esthetic score | Pink esthetics will be measured using pink esthetic index chart After 6 months.
  Will be measured using pink esthetic index chart

IPD SHARING:
Plan to Share IPD: Undecided